CLINICAL TRIAL: NCT00056290
Title: p.VGI.1 (VEGF2) Gene Transfer for Diabetic Neuropathy
Brief Title: VEGF Gene Transfer for Diabetic Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Losordo, Douglas, M.D. (Individual)
Responsible Party: Director, Feinberg Cardiovascular Research Institute, Program in Cardiovascular Regenerative Medicine, Northwestern University, Northwestern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BB-IND 11572; NIH #0104-467
Expanded Access: Available
Record Dates: First submitted 2003-03-10; First posted 2003-03-11 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetes Mellitus; Neuropathy; Peripheral Artery Disease
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Peripheral Arterial Disease | interventions — Vascular Endothelial Growth Factor A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): VEGF
  Interventions: Biological: VEGF
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: VEGF

INTERVENTIONS:
Biological: VEGF — 3 sets of injections, at 2 week intervals
  Arms: 1
Biological: VEGF — 3 sets of injections, at 2 week intervals
  Arms: 2

SUMMARY:
This gene therapy study is being conducted to evaluate intramuscular gene transfer using VEGF (Vascular Endothelial Growth Factor) in patients with diabetic neuropathy in the legs. This condition causes a decrease in feeling and sensation due to diabetes. VEGF is DNA, or genetic material that is injected into the muscles of the leg. Once in the leg, it has been shown to cause new blood vessels to grow under a variety of conditions.

ELIGIBILITY:
Inclusion criteria:

To be eligible to enroll and remain in the study, patients must meet the following criteria:

* Be at least 21 years old.
* Have type I or type II diabetes mellitus and require oral anti-hyperglycemic agents or insulin.
* Have peripheral neuropathy related to diabetes.

Exclusion criteria

Patients are to be excluded from the trial if any of the following conditions are met:

* Have a history of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Be unable to meet study requirements, including approximately 7-9 out-patient visits over a 12 month period.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2002-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Safety | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan H Ropper, M.D., Principal Investigator — Steward St. Elizabeth's Medical Center of Boston, Inc.
Locations (2):
- United States (2):
  - Caritas St. Elizabeth's Medical Center Cardiovascular Research/DVM-4-SMC, Boston, Massachusetts
  - Columbia University Neuropathy Research Center, Neurological Institute, New York, New York

REFERENCES:
- See also: Caritas St. Elizabeth's Medical Center of Boston — http://www.semc.org